CLINICAL TRIAL: NCT04636177
Title: Pain Rehabilitation Virtual Reality (PRVR): Innovations to Enhance Mobility in the Presence of Pain
Acronym: PRVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Laura E Simons, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68669; R21AR079140 (NIH)
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Fibromyalgia; Virtual Reality
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Rehabilitation Virtual Reality (PRVR) (Experimental): Participants will complete VR in PT to engage participants in a series of immersive games customized to align with individual PT needs delivered over ~6-12 weeks or until clinician believes the patient is done with treatment. Patients in the PRVR arm will be given a structured HEP to practice prescribed exercises at home with integrated VR activities. PRVR participants will be allocated a VR headset for use in PT sessions and with HEP. VR will supplement treatment and be used in session (either in-person or telehealth) and at home as part of their prescribed treatment homework.
  Interventions: Behavioral: Pain Rehabilitation Virtual Reality (PRVR)
- Standard Physiotherapy Rehabilitation (SPR) (Active Comparator): Sessions are individually-tailored and based on the Guide to Physical Therapy Practice 3.0 consisting of 1) therapeutic exercise, 2) balance and proprioception, 3) strength training, and 4) use of modalities (e.g., heat/cold pack). Patients will be given a structured Home Exercise Program (HEP) with prescribed exercises for home. SPR participants will be allocated a VR headset for recreational use.
  Interventions: Behavioral: Standard Physiotherapy Rehabilitation (SPR)

INTERVENTIONS:
Behavioral: Pain Rehabilitation Virtual Reality (PRVR) — Participants will receive approximately 8, 1-hour physiotherapy sessions delivered over the course of 6-12 weeks. Adequate dose: 75% (6 of 8 sessions).
  Arms: Pain Rehabilitation Virtual Reality (PRVR)
Behavioral: Standard Physiotherapy Rehabilitation (SPR) — Participants allocated to either intervention arm will receive 8, 1-hour physiotherapy sessions delivered over the course of 6-8 weeks. Adequate dose: 75% (6 of 8 sessions).
  Arms: Standard Physiotherapy Rehabilitation (SPR)

SUMMARY:
The proposed research is a single arm feasibility trial of pain rehabilitation virtual reality (PRVR) aimed at measuring feasibility, acceptability and utility of VR as well as changes in physical function and fear for adolescents with chronic musculoskeletal pain. The intervention includes standard physiotherapy treatment including functional goal setting and progressive exercise.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 17 years old
* Musculoskeletal pain (e.g. localized [back, limb], diffuse) not due to acute trauma (e.g. active sprain or fracture)
* English Language Proficiency

Exclusion Criteria:

* Significant cognitive impairment (e.g., brain injury)
* Significant medical or psychiatric problem that would interfere (e.g. psychosis, suicidality)
* Presents with a condition that interferes with virtual reality usage (e.g., history of seizure, facial injury precluding safe placement of headset, visual impairment, significant hearing impairment impact ability to follow audio instructions).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Simons, PhD, Principal Investigator — Stanford School of Medicine
Locations (2):
- United States (2):
  - Pediatric Pain Management Clinic - Stanford Children's Health, Menlo Park, California
  - California Rehabilitation and Sports Therapy, Palo Alto, California

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (text, tables, figures, appendices) that underlie the results reported in an article related to this trial will, after de-identification, be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to Dr. Laura Simons at lesimons@stanford.edu. To gain access, data requestors will need to sign a data access agreement with Stanford University.

REFERENCES:
- [Derived] Simons LE, Hess CW, Choate ES, Van Orden AR, Tremblay-McGaw AG, Menendez M, Boothroyd DB, Parvathinathan G, Griffin A, Caruso TJ, Stinson J, Weisman A, Liu T, Koeppen K. Virtual Reality-Augmented Physiotherapy for Chronic Pain in Youth: Protocol for a Randomized Controlled Trial Enhanced With a Single-Case Experimental Design. JMIR Res Protoc. 2022 Dec 12;11(12):e40705. doi: 10.2196/40705. PMID 36508251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was originally conceived as a two-arm study, with patients randomized 1:1 to Pain Rehabilitation Virtual Reality (PRVR) or Standard Physiotherapy Rehabilitation (SPR). Early in the study, the design was changed from that point all participants were allocated to the PRVR arm.
Groups:
- Pain Rehabilitation Virtual Reality (PRVR): PRVR participants are allocated a VR headset for use in their physical therapy sessions and as part of their home exercise program (approximately 8, 1-hour physiotherapy sessions delivered over the course of 6-12 weeks).
- Standard Physiotherapy Rehabilitation (SPR): SPR participants are allocated to sessions that are individually-tailored and based on the Guide to Physical Therapy Practice 3.0 as part of their home exercise program (8, 1-hour physiotherapy sessions delivered over the course of 6-8 weeks).
Period: Two-arm, randomization portion
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Started | 4 | 6
Completed | 3 | 4
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Single-arm portion
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Started (All participants starting this period were new) | 24 | 0
Completed | 22 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR) | Total
Number analyzed (Participants) | 28 | 6 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 6 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 14 | 0 | 14
  Other | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 25 | 5 | 30
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 0 | 1 | 1
  White | 16 | 3 | 19
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 6 | 34

OUTCOME MEASURES:

1. Primary Outcome: VR Duration of Use Per Week
Description: This outcome is to assess Feasibility, Acceptability, and Utility of VR.
Time Frame: Baseline to end of treatment across 6-8 weeks, on average
Population: Participants who completed the protocol
Measure: Mean (Standard Deviation); unit: Minutes per week
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Number analyzed (Participants) | 25 | 4
Minutes per week | 30.5 (39.52) | 17.0 (6.36)

2. Primary Outcome: Participant Rated Ease of Use
Description: This outcome is to assess Feasibility, Acceptability, and Utility of VR.
Time Frame: End of treatment at 6-8 weeks, on average
Population: Participants who completed the protocol
Measure: Count of Participants; unit: Participants
Groups:
- Standard Physiotherapy Rehabilitation (SPR): SPR participants are allocated to sessions that are individually-tailored and based on the Guide to Physical Therapy Practice 3.0 as part of their home exercise program (8, 1-hour physiotherapy sessions delivered over the course of 6-8 weeks). Participants receive standard VR headset with relaxing games.
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Number analyzed (Participants) | 25 | 4
Participants
  Very easy | 13 | 0
  Easy | 6 | 3
  A little easy | 4 | 0
  Not at all easy | 0 | 0
  No Response | 2 | 1

3. Primary Outcome: Participant Rated Enjoyment
Description: This outcome is to assess Feasibility, Acceptability, and Utility of VR.
Time Frame: End of treatment at 6-8 weeks, on average
Population: Participants who completed the protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Number analyzed (Participants) | 25 | 4
Participants
  Enjoyed very much | 5 | 0
  Enjoyed | 10 | 0
  Enjoyed a little | 5 | 3
  Not at all | 0 | 0
  No response | 5 | 1

4. Secondary Outcome: Pain-related Fear and Avoidance
Description: Fear of Pain Questionnaire Short Form (FOPQ- SF): a 10-item validated patient-reported measure of pain-related fear and avoidance. Total score range: Min=0, Max=40; lower score indicates less fear and avoidance/better outcomes.
Time Frame: Baseline to end of treatment at 6-8 weeks, on average and at 3-months after end of treatment
Population: Participants who were enrolled in the study were analyzed at baseline and those who completed treatment and 3-month follow-up surveys were analyzed at those timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Number analyzed (Participants) | 28 | 6
score on a scale
  baseline | 21.00 (8.67) | 18.00 (3.41)
  end of treatment: number analyzed (Participants) | 25 | 4
  end of treatment | 15.84 (9.66) | 17.5 (11.7)
  3-month follow-up: number analyzed (Participants) | 25 | 4
  3-month follow-up | 15.58 (8.05) | 22.00 (13.64)

5. Secondary Outcome: Physical Function: Lower Extremity
Description: Lower Extremity Functional Scale (LEFS): a 20-item validated patient-reported measure of lower extremity function. Overall score range: Min=0, Max=80; lower score indicates greater disability/worse outcomes.
Time Frame: Baseline to end of treatment at 6-8 weeks, on average and at 3-months after end of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Number analyzed (Participants) | 28 | 6
score on a scale
  baseline | 54.64 (14.13) | 46.83 (19.90)
  end of treatment: number analyzed (Participants) | 25 | 4
  end of treatment | 63.24 (11.57) | 57.75 (16.64)
  3-month follow-up: number analyzed (Participants) | 25 | 4
  3-month follow-up | 66.76 (11.73) | 71.50 (9.57)

6. Secondary Outcome: Physical Function: Upper Extremity
Description: Upper Extremity Functional Index (UEFI): a 20- item validated patient-reported measures of upper extremity functioning. Overall score range: 0 to 80, with greater scores indicating increased upper extremity functioning.
Time Frame: Baseline to end of treatment at 6-8 weeks, on average and at 3-months after end of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
Number analyzed (Participants) | 28 | 6
score on a scale
  baseline | 64.07 (12.84) | 69.83 (14.61)
  end of treatment: number analyzed (Participants) | 25 | 4
  end of treatment | 67.48 (10.42) | 75.75 (3.5)
  3-month follow-up: number analyzed (Participants) | 25 | 4
  3-month follow-up | 72.40 (7.96) | 78.00 (3.37)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Pain Rehabilitation Virtual Reality (PRVR) | Standard Physiotherapy Rehabilitation (SPR)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/6
Other Adverse Events (participants affected / at risk) | 1/28 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pain Rehabilitation Virtual Reality (PRVR) (N=28) | Standard Physiotherapy Rehabilitation (SPR) (N=6)
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT04636177/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT04636177/ICF_002.pdf